CLINICAL TRIAL: NCT00844870
Title: Training With or Without Upper Body Restraint During Reaching in Individuals Post Stroke
Brief Title: Exploring New Approaches in Reaching Behavior Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Sciences in Philadelphia (Other)
Responsible Party: Gregory Thielman, University of The Sciences in Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-007
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Stroke
Keywords: rehabilitation, reaching, stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): stabilization training group
  Interventions: Behavioral: stabilization training
- 2 (Experimental): auditory response training group
  Interventions: Behavioral: auditory training group

INTERVENTIONS:
Behavioral: stabilization training — training of arm function with the trunk stabilized
  Arms: 1
Behavioral: auditory training group — response to an auditory signal
  Arms: 2

SUMMARY:
After 4 weeks of training the hypothesis that the more natural training program would yield greater functional changes was proven correct.

DETAILED DESCRIPTION:
Analysis indicated that both methods improved reaching without trunk use Reaching performance scale (RPS), but the trunk -stabilized group led to more significant changes. Training under less restrictive conditions associated with Task-Related Training (TRT) (auditory feedback from trunk sensor) as compared to stabilized TRT, led to improved functional and impairment measure scores (WMFT, FM and shoulder flexion). Conclusion: Fading feedback with both training methods, during extended TRT reaching/grasping practice generally led to some improvements. However, as demonstrated by impairment and functional outcome measures, using TRT with an auditory feedback signals is a more effective approach than forcing the stabilization of the trunk during rehabilitation of the upper-limb.

ELIGIBILITY:
Inclusion Criteria:

* Individuals all scored between 20 and 44 on the Upper-Arm subsection of the Fugl-Meyer Scale (FM- Poole & Whitney, 1988) and demonstrated some trunk movement during the pretest reaching performance scale measures (RPS, Levin 2006)

Exclusion Criteria:

* Individuals were referred if they had no receptive aphasia, apraxia or other cognitive deficits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
WMFT | 1 year

SECONDARY OUTCOMES:
FM and shoulder flexion | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gregory T Thielman, Ed.D, Principal Investigator — University of the Sciences in Philadelphia